CLINICAL TRIAL: NCT00487838
Title: Noninvasive Optical Imaging of the Effects of External Spectral Filters on Macular Autofluorescence in Pseudophakic Eyes
Brief Title: Effects of Sun Filters on Age-related Macular Degeneration in People With Lens Implants
Status: Withdrawn | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070169; 07-CH-0169
Record Dates: First submitted 2007-06-16; First posted 2007-06-19 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-05-04

CONDITIONS: Age-Related Macular Changes; Age-Related Macular Degeneration; Cataract and IOL Surgery; Retinal Photochemistry
Keywords: Autofluorescence Imaging; Early Age-Related Maculopathy; Photochemical Changes; Colored Sunglasses; Pseudophakes; Fundus Camera; Confocal Scanning Laser Ophthalmoscope; Molecular Imaging within Retina; Spectral Balance among Photochemical Processes; Noninvasive Autofluorescence Imaging; Age-Related Maculopathy (AMD); Age-Related Macular Degeneration; AMD; Age-Related Macular Changes; Early Age-Related Macular Changes
MeSH Terms: conditions — Macular Degeneration; Cataract

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will test a new method for preventing worsening of age-related macular degeneration (AMD) and for developing imaging methods to follow the very earliest microscopic changes in the disease. The macula is the part of the retina in the back of the eye that determines central vision. AMD can impair central vision, affecting a person's ability to read, drive, and carry out daily activities. Some studies suggest that cumulative exposure to sunlight increases the risk for progression of AMD to the late stage that is often characterized by poor central vision. This study will determine if wearing glasses with a yellow filter over one eye and a red-violet filter over the other eye when outdoors will decrease the rate of change of early-stage AMD in one or both eyes.

Patients early-stage AMD who have had cataract surgery in both eyes with implanted lenses may be eligible for this study.

Participants undergo the following procedures:

* Wear the filter glasses when outdoors between 10:00 a.m. and 4:00 p.m.
* Record the time of day and light environment when they use the glasses.
* Have an eye examination, pictures of the retina, and a medical history taken at the beginning of the study and at set intervals during the study.

The study lasts at least 12 months and may be extended for a longer period of time....

DETAILED DESCRIPTION:
Accumulation of the photoproduct N-retinylidene-n-retinylethaholamine (A2E) within the retina may be associated with the early age-related macular degeneration (AMD). Our biophysical model of retinal photochemistries predicts that as the lens yellows with age a spectral imbalance of the light reaching the retina causes steady-state A2E levels to rise in the RPE, which induces increasing RPE stress leading to AMD progression. If correct, this rise in A2E levels and the initial injury could be prevented by appropriately chosen spectral filtering (e.g., colored sunglasses). Autofluorescence imaging of the retina currently allows noninvasive mapping of total accumulated lipofuscin fluorophores within the macular retinal pigment epithelium (RPE) but not A2E or its precursor alone. By adding new sets of excitation and emission filters to existing fundus cameras and confocal scanning laser ophthalmoscopes, we propose to map individually both A2E and its precursor A2PEH2 or their fractional contributions to the total retinal fluorescence. By following A2E fluorescence in both eyes in subjects following bilateral cataract surgery and intra-ocular lens [IOL] implantation with early symmetric age-related maculopathy who wear our bicolored sunglasses whenever outdoors in the daylight, we propose to test this hypothesis while efficiently controlling for hidden genetic, physiological, and environmental confounding variables between subjects. This pilot protocol seeks to optimize recruitment of suitable subjects and the reproducibility of our spectral imaging and noninvasive analysis of A2E and A2PEH2 levels in the normal and microscopically abnormal regions of the macula. The data from this pilot study will be used to design a clinical study to test our hypothesis.

ELIGIBILITY:
* INCLUSION CRITERIA:

All eligible patients are invited to participate in this study.

Patients will be local area residents who average greater than or equal to 2 hours outdoors daily, who are willing to follow the protocol of wearing our bicolor sunglasses whenever outdoors in daylight and to keep a log book of use and to return periodically to NIH for our noninvasive imaging studies.

EXCLUSION CRITERIA:

Individuals with signs of more advanced age-related maculopathy in either eye such as identifiable regions of geographic atrophy or choroidal neovascularization.

Individuals with prior eye disorders (other than uncomplicated cataract surgery and early age-related maculopathy).

Individuals with diabetes mellitus, current chemotherapy, or other medicines or conditions that may affect our ability to perform accurate autofluorescence imaging or interfere with follow-up visits.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-06-14; Study Completion 2012-05-04

CONTACTS AND LOCATIONS:
Overall Officials: Jack A Yanovski, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)

REFERENCES:
- [Background] Klein R, Klein BE, Linton KL. Prevalence of age-related maculopathy. The Beaver Dam Eye Study. Ophthalmology. 1992 Jun;99(6):933-43. doi: 10.1016/s0161-6420(92)31871-8. PMID 1630784
- [Background] Taylor HR, West S, Munoz B, Rosenthal FS, Bressler SB, Bressler NM. The long-term effects of visible light on the eye. Arch Ophthalmol. 1992 Jan;110(1):99-104. doi: 10.1001/archopht.1992.01080130101035. PMID 1731731
- [Background] Tomany SC, Cruickshanks KJ, Klein R, Klein BE, Knudtson MD. Sunlight and the 10-year incidence of age-related maculopathy: the Beaver Dam Eye Study. Arch Ophthalmol. 2004 May;122(5):750-7. doi: 10.1001/archopht.122.5.750. PMID 15136324